CLINICAL TRIAL: NCT01476618
Title: Providing Mental Health Services to Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans: Provider Perspectives
Brief Title: Providing Mental Health Services to Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gina Signoracci, Psychology Post-Doctoral Fellow, VA Eastern Colorado Health Care System
Other Study IDs: 11-0300
Record Dates: First submitted 2011-11-07; First posted 2011-11-22 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Mental Health Services
Keywords: Provider Perspectives; Barriers; OIF/OEF Veterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Denver VA OIF/OEF and mental health providers: Denver VA OIF/OEF and mental health providers
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to gather information from VISN 19 Denver VA mental health professionals regarding their perspectives of necessary resources to provide best practice mental health service to Operation Iraqi Freedom (OIF)/ Operation Enduring Freedom (OEF) Veterans. Specifically, this study aims to describe provider perspectives regarding the following: a) clinical needs of OIF/OEF Veterans; b) collaboration and referral processes; c) barriers to providing optimal treatment to this cohort d) provider needs and resources that may improve service delivery to this cohort; e) provider perspectives regarding psychiatric outcomes in this cohort; and f) professional satisfaction. Support for this study is provided by previous research evaluating Veteran's Administration (VA) needs to provide service to OIF/OEF Veterans (Sayer, et al. 2009; Friedmann-Sanchez, et al. 2008).

The above information will be obtained using semi-structured interview. Hypotheses are not provided as this is an exploratory qualitative study.

DETAILED DESCRIPTION:
No hypotheses are associated with this study as this is a qualitative study wherein subjects will participate in a semi-structured interview developed specifically for this study, which serves as the outcome measure. Up to 30 providers will be interviewed.

Data Analysis Interviews will be transcribed in their entirety and de-identified. Dr. Signoracci and 4 additional MRIECC researchers will independently code each interview for themes. Finally, group meetings with Dr. Signoracci and MIRECC researchers will be held in order to achieve larger consensus regarding such unique and universal themes (Rubin & Rubin, 1995).

Any reporting of information regarding: a) length of time employed at Denver VA; b) length of time employed within VA system; c) provider professional title; d) provider degree; f) professional licenses held; g) clinic/service in which provide services will be done in the aggregate, across clinics. No individual data will be reported with respect to these items. Also, any selected quotes that are reported will remain de-identified.

Power analyses will not be conducted because no hypothesis quantitative testing is being done, and therefore there are no parameters to estimate. With qualitative designs one conducts interviews until reaching the saturation point. In other words, subsequent interviews do not yield any new information (Rubin & Rubin, 1995). Previous experience (Brenner et al., 2008) suggests that 25 completed interviews should provide a wide enough range of responses for important themes to emerge.

ELIGIBILITY:
Inclusion Criteria

* Denver VA Mental Health Providers that provide mental health treatment to OIF/OEF Veterans
* Age 18-70

Exclusion Criteria Denver VA providers that do not provide mental health to OIF/OEF Veterans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Denver VA Mental Health Providers Up to 30 providers will be interviewed.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interview | Interview conducted one time per participant (completion time: approximately 1 hour)
  Semi-structured interview regarding provider experiences of providing mental health treatment to OIF/OEF Veterans. The interview takes approximately 1 hour to complete and is conducted one time with each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Gina M Signoracci, Ph.D., Principal Investigator — VISN 19 Denver VA MIRECC
Locations (1):
- Denver VA, Denver, Colorado, United States